CLINICAL TRIAL: NCT00734045
Title: Prospective Evaluation of the StatusFirst™ CHF NT-proBNP Device in Human Whole Blood and Plasma Samples
Acronym: WB-13
Status: Completed | Type: Observational
Sponsor: Nanogen, Inc. (Industry)
Responsible Party: Philip Estes / Associate Director, Clinical, Nanogen
Other Study IDs: WB-13
Record Dates: First submitted 2008-08-11; First posted 2008-08-13 (Estimated); Last update posted 2008-12-10 (Estimated); Status verified 2008-12

CONDITIONS: Congestive Heart Failure (CHF)
Keywords: Congestive Heart Failure (CHF); NT-proBNP
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Subjects with diagnosed congestive heart failure
- 2: Subjects not diagnosed with congestive heart failure

SUMMARY:
The primary objective of the study is to establish the correlation between NT-proBNP measurements in fresh human whole blood samples and those in plasma samples from the same study subjects, where said samples are collected in EDTA and Li-Hep anticoagulant tubes and measured by the StatusFirst™ CHF NT-proBNP device in conjunction with the DXpressTM Reader in a laboratory setting.

ELIGIBILITY:
Inclusion Criteria:

* Have clinically confirmed heart failure (NYHA class I-IV) or have presented to an emergency room or clinic with signs, symptoms and/or risk factors suggestive of heart failure, OR
* Be non-CHF controls greater than 45 years of age with no history of heart failure or cardiovascular disease.

Exclusion Criteria:

* Be 45 years of age or younger

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients to be recruited for the study should either:
  * have clinically confirmed heart failure (NYHA class I-IV) or have presented to an emergency room or clinic with signs, symptoms and/or risk factors suggestive of heart failure, OR
  * be non-CHF controls greater than 45 years of age with no history of heart failure or cardiovascular disease.
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2008-02; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
StatusFirst CHF NT-proBNP test result | At presentation to study site (no follow-up)

CONTACTS AND LOCATIONS:
Overall Officials: Alan Wu, PhD, Principal Investigator — University of California San Francisco and San Francisco General Hospital; Alan Maisel, MD, Principal Investigator — University of California San Diego; Veteran's Affairs
Locations (2):
- United States (2):
  - US Department of Veteran's Affairs, San Diego, California
  - San Francisco General Hospital, San Francisco, California